CLINICAL TRIAL: NCT03489681
Title: Acupuncture Treatment on Chronic Sciatica: the Efficacy, Mechanism, and Functional Neuroimaging Pain-network Study
Brief Title: Acupuncture Treatment for Chronic Sciatica: the Neuroimaging Pain-network Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: Lotung Poh-Ai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-01-014A
Record Dates: First submitted 2017-12-21; First posted 2018-04-05 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Therapy, Acupuncture; MRI, Functional
Keywords: acupuncture, sciatica, default mode network
MeSH Terms: conditions — Sciatica | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: The investigators performed a prospective, randomized controlled study with three arms, the high-dose acupuncture, low-dose acupuncture, and healthy controlled groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupuncture, low dosage (Experimental): treat as six acupoints
  Interventions: Device: acupuncture
- Acupuncture, high dosage (Experimental): treat as 18 acupoints
  Interventions: Device: acupuncture
- Control group (No Intervention): no acupuncture treatment, healthy control

INTERVENTIONS:
Device: acupuncture — Low dose group:
  Twenty patients will assign for low dose group treatment; as six acupoints as Shensu (BL 54), Huantiao (GB 30), Weizhong (BL 40), Yanglingquan (GB 34), Kunlun (BL 60), Juegu (GB 39).
  High dose group:
  Twenty patients will assign for high dose group treatment. These acupoints contains of eighteen acupoints, as Shenshu (BL 54), Dachangshu (BL 25) , Xiaochangshu (BL 27), Huantiao (GB 30), Yinmen (BL 37) , Zhibien (BL 54), Chengfu (BL 36), Fengshi (GB 31), Weizhong (BL 40), Zusanli (ST 36) Yanglingquan (GB 34), Yinlingquan (SP 9), Feiyang (BL 58), Sanyinjiao (SP 6), Juegu (GB 39), KunLun (BL 60), , Taixi (KI 3), Shenmai (BL 62).
  Other Names: Ching Ming Mdical Device Co, Taipei, Taiwan, R.O.C
  Arms: Acupuncture, high dosage; Acupuncture, low dosage

SUMMARY:
Sciatica is a common pain disorder in the neurological clinic that typically present as low back or gluteal pain and may radiate to one leg with motor or sensory complaint. Sciatica has drawn more attention worldwide as a public health issue for its pain disability, high prevalence and significant medical and economic burden. A meta-analysis of sciatica treatment revealed discectomy, epidural injections, non-opioid analgesics, and acupuncture might relieve pain. However, the central effect of acupuncture-induced analgesia and its functional connectivities in various brain region remain unclear. Besides, the number of acupoints selection and its correlation in functional connectivity also need to be discussed. This clinical trial would collect the sciatica subjects assign by intent to treat, divided to acupuncture and non-acupuncture herbal control group. The treatment of acupuncture assigns randomized as high dose and low dose acupuncture group. The acupuncture will perform two times a week for four weeks. The primary outcomes are visual analog scale for pain and sciatica bothersomeness index; the secondary outcomes are Roland's disability questionnaire for sciatica, WHOQOL, and traditional Chinese medical constitutional scale. The functional magnetic resonance imaging scan would apply at the baseline and after four weeks' treatment. This study aims to explore the model of DMN in sciatica patients; it's central effect in different stimulation modality and to investigate the mechanism of the long-lasting, sustained impact in different acupuncture dosage.

ELIGIBILITY:
Inclusion Criteria:

1. 35 - 70 y/o.
2. Low back or gluteal pain radiating into one leg.
3. Pain duration of at least two weeks.

Exclusion Criteria:

1. Known or suspected severe spinal pathology (for example, cauda equina syndrome, or spinal fracture).
2. Pregnant or breastfeeding women.
3. Scheduled or being considered for spinal surgery or interventional procedures for sciatica during the 8-week treatment period.
4. Administration of sedative or analgesics within 24 h before the fMRI scan.
5. Comorbidities include systemic malignancy, bleeding tendency, rheumatic arthritis and other known autoimmune diseases.
6. Focal neurologic deficits with progressive or disabling symptoms
7. History of received acupuncture treatment in the past one month.
8. Any contraindication related to acupuncture and MRI.
9. Visual analog scale < 3.
10. Low back pain without sciatica.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Change from Baseline VAS at 4 weeks
  pain scale; from 0 to 10; score 0: no pain, score 10: unbearable pain, the higher values represent, the worse outcome

SECONDARY OUTCOMES:
Sciatica Bothersome Index (SBI) | Change from Baseline SBI at 4 weeks
  score 0: not bothersome; score 24: extremely bothersome, the higher values represent, the worse outcome
Roland Disability Questionnaire for Sciatica (RDQS) | Change from Baseline RDQS at 4 weeks
  Evaluation of Disability of sciatica; score 0: not the disability, score 24: most disability; the higher values represent, the worse outcome
The World Health Organization Quality of Life -brief edition (WHOQOL-Brief) | Change from Baseline WHOQOL-Brief at 4 weeks
  evaluation of daily life quality; the more the scores, the better the quality of life subscale: 1 Physical health (score 4-20); 2 Psychological (score 4-20); 3 Social relationships(score 4-20); 4 Environment (score 4- 20), total score: minimum 8, maximum 80); the higher values represent, the better outcome
Body Constitution Questionnaire (BCQ) | baseline (1st time rsMRI examination)
  Traditional Chinese medicine (TCM), is an ancient system of personalized medicine based on body constitution (BC) theory. BC is the fundamental physiological component of a person, and different BC types are variously susceptible to disease and affect the development and prognosis of diseases. Patient classification is important in TCM, Body Constitution Questionnaire (BCQ) is developed by Prof. Su (Taiwan,2009); which classified people with their personalized trait 'body constitution' and scoring as 'Yin- deficiency', Yang-deficiency' and 'Phlegm & dampness'. The more the scores, the more tendency of the BCQ sub-type( cut off point, 30 points, 31 points, and 27 points respectively).

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Liu CH, Kung YY, Lin CL, Yang JL, Wu TP, Lin HC, Chang YK, Chang CM, Chen FP. Therapeutic Efficacy and the Impact of the "Dose" Effect of Acupuncture to Treat Sciatica: A Randomized Controlled Pilot Study. J Pain Res. 2019 Dec 31;12:3511-3520. doi: 10.2147/JPR.S210672. eCollection 2019. PMID 32021387